CLINICAL TRIAL: NCT02730923
Title: A Multicentric, Randomized, Non Comparative, Open-label Phase I/II Evaluating AZD2014 (Dual Mammalian Target of Rapamycin Complex 1/2 (mTORC1/mTORC2) Inhibitor) in Combination With Anastrozole Versus Anastrozole Alone in the Treatment of Metastatic Hormone Receptor-positive Endometrial Adenocarcinoma
Brief Title: Hormone Receptor Positive endometrIal Carcinoma Treated by Dual mTORC1/mTORC2 Inhibitor and Anastrozole (VICTORIA)
Acronym: VICTORIA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICTORIA (ET150036)
Record Dates: First submitted 2016-03-18; First posted 2016-04-07 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2023-09

CONDITIONS: Endometrial Carcinoma; Metastatic Carcinoma; Hormone Receptor Positive Tumor
Keywords: Clinical Trials, Randomized; Clinical Trial, Phase I; Clinical Trial, Phase II; Multicenter Trials; Aromatase Inhibitors; mTOR kinase inhibitor
MeSH Terms: conditions — Endometrial Neoplasms; Carcinoma | interventions — vistusertib; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: AZD2014 plus anastrozole (Experimental)
  Interventions: Drug: AZD2014; Drug: Anastrozole
- Arm B: anastrozole alone (Active Comparator)
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: AZD2014 — Following inclusion, patients will be randomized (2:1) to receive Arm A : AZD2014 + anastrozole Arm B : anastrozole alone
  Mode of Action Selective and specific mTOR kinase inhibitor targeting both mTORC1 and mTORC2 complexes.
  Route of Administration Oral
  Dosage regimen 125mg BID with intermittent schedule (2 days of treatment followed by 5 days off (500mg/week))
  Duration of treatment Until the patient experiences unacceptable toxicity, disease progression and/or treatment is discontinued per patient or investigator request.
  Arms: Arm A: AZD2014 plus anastrozole
Drug: Anastrozole — Therapeutic Class Aromatase inhibitor
  Mode of Action Potent and highly selective non-steroidal aromatase inhibitor.
  Route of Administration Oral
  Dosage regimen
  1 mg tablet once a day
  Duration of treatment Patients may continue treatment with anastrozole until the patient experiences unacceptable toxicity, disease progression and/or treatment is discontinued per patient or investigator request.
  Other Names: Arimidex

SUMMARY:
The investigators hypothesize that the dual inhibition of mTORC1/mTORC2 by AZD2014 combined with inhibition of aromatase enzyme by anastrozole will act synergistically and may be an interesting therapeutic option for endometrial cancer with a manageable toxicity profile.

The investigators proposal is to conduct a multicenter, 2-step, randomized, Phase I/II trial to evaluate the safety and efficacy of a combination treatment associating anastrozole to AZD2014 in advanced endometrial cancer patients.

The study is divided in 2 steps :

* A safety run-in phase aiming to evaluate the safety of the proposed combination AZD2014 + anastrozole (Arm A) versus anastrozole alone (Arm B). No dose escalation is scheduled (doses are based on maximum tolerated dose (MTD) defined for AZD2014 and the summary of product characteristics (SPC) of anastrozole). However, dose de-escalation for AZD2014 will be applied in case of toxicity.
* A two-stage randomized Phase II part aiming to evaluate the clinical benefit of the AZD2014 + anastrozole (Arm A) combination therapy versus anastrozole (Arm B).

DETAILED DESCRIPTION:
TREATMENT PLAN :

Following randomisation patients will receive Arm A : AZD2014 plus anastrozole or Arm B: anastrozole alone AZD2014 will be administered with an intermittent schedule i.e. 125 mg bis in die (BID) intermittent with 2 days on followed by 5 days off per week for a total weekly dose of 500 mg/week (250mg D1 and D2, 5 days off) Anastrozole will be administered at the standard dose defined in the SPC i.e. 1mg/d, per os, continuously.

Both treatment will be administered until progressive disease (PD), unacceptable toxicity or willingness to stop.

STATISTICS :

A total of 72 patients will be randomized in the study.

Safety run-in Phase on the first 9 patients randomized - As no dose escalation will be performed, the safety will be evaluated following the treatment and 8-week follow-up of the first 6 patients by the experimental association AZD2014+anastrozole (experimental arm). By similarity to a classic 3+3 design, based on binomial probabilities, there is a 90% probability of observing one or more patients with a toxicity event, if that event occurs in at least 32% of the target population. Assuming a 2:1 randomization ratio, a total of 9 patients (Arm A - Experimental: 6 patients, Arm B - Control: 3 patients) will be enrolled in this safety run-in phase and will be included in the evaluation of Phase II part.

Phase II The sample size calculation was based on a Simon optimal two-stage design, with a minimum success (8-week non progression) rate considered of interest p1=60% and an uninteresting rate p0=40%. Assuming a type I error alpha of 0.05 and 80% power, 46 evaluable patients are needed in the experimental arm to reject the null hypothesis H0: p≤p0 versus the alternative hypothesis H1: p ≥ p1 in a unilateral situation (16 patients in Stage I and 30 additional patients in Stage II).

With a 2:1 randomization and based on the assumption that 5% of the patients may be non-evaluable, a total of 72 patients will be included in the study : 48 patients in Arm A - experimental and 24 patients in Arm B - control).

DATA ENTRY, DATA MANAGEMENT AND STUDY MONITORING All the data concerning the patients will be recorded in the electronic case report form (eCRF) throughout the study. serious adverse event (SAE) reporting will be also paper-based by e-mail and/or Fax.

The sponsor will perform the study monitoring and will help the investigators to conduct the study in compliance with the clinical trial protocol, Good Clinical Practices (GCP) and local law requirements.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female patient at the time of consent
* Histologically-confirmed diagnosis of advanced or recurrent endometrial carcinoma, not amenable to curative treatments. Carcinosarcoma are not eligible.
* Documented estrogen receptor and/or progesterone receptor positive endometrial cancer. Hormone receptor positivity is defined according to routine practice at each participating site.
* Availability of a pre-treatment tumor sample (archival formalin-fixed paraffin-embedded (FFPE) block or fresh biopsy if feasible) and presence of at least one biopsiable tumor lesion for on-treatment biopsy
* Documented disease progression after no more than one prior first-line chemotherapy regimen and/or more than 2 lines endocrine therapy in the metastatic setting
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1 and minimum life expectancy of 8 weeks
* At least one measurable lesion according to response evaluation criteria in solid tumor (RECIST 1.1)
* Adequate bone marrow, renal and liver function as shown by:

  * Absolute neutrophil count > 1.5 x 109/L, Platelets > 100 x 109/L, Hemoglobin (Hb) >9 g/dL
  * Serum bilirubin ≤ 1.5 upper limit of normal (ULN), alanine aminotransferase and aspartate aminotransferase ≤ 2.5 ULN (≤ 5 ULN in patients with liver metastases)
  * Creatinine clearance > 50 mL/min (using Cockcroft formula, or MDRD formula for patients over 65 years Appendix 3 - Creatinine Clearance)
* Fasting serum cholesterol ≤ 300 mg/dL (7.75 mmol/L) AND fasting triglycerides ≤ 2.5 ULN (lipid-lowering drugs allowed),
* Fasting plasma glucose ≤7 mmol/L (126 mg/dL)
* Recovered from prior significant treatment-related toxicity i.e. no persistent treatment-related toxicity > Grade 1 as per Common Terminology Criteria for Adverse Events (CTCAE) v4.3, except grade 2 alopecia, grade 2 anemia but with Hb >9 g/dL.
* Minimal wash-out period before the start of the study drugs for the following treatments:

  * Any anti-cancer treatment approved or investigational medicinal product :> 21 days
  * Any chemotherapy, radiation therapy, androgens : > 21 days (not including palliative radiotherapy at focal sites).
  * Any monoclonal antibody therapy: > 4 weeks
  * Major surgery: > 4 weeks
  * Minor surgery (excluding tumour biopsies) >14 days.
  * Any haemopoietic growth factors (e.g., filgrastim [granulocyte colony-stimulating factor (G-CSF)], sargramostim [granulocyte-macrophage colony-stimulating factor (GM-CSF)]): > 14 days
  * Vaccinated with live, attenuated vaccines : > 4 weeks.
* Sensitive or narrow therapeutic range substrates of drug transporters OATP1B1, OATP1B3, MATE1 and MATE2K: see the appropriate wash-out period (a minimum of 5 x reported elimination half-life) in Appendix 5 - Restricted CYP and transporter related co-medications
* Potent or moderate inhibitors or inducers of CYP3A4/5, Pgp (MDR1) and BCRP - Restricted CYP and transporter related co-medications
* Patient willing to follow sunlight-protection measures. Patients should be advised of the need for sunlight protection measures during administration of AZD2014, and should be advised to adopt such measures for a period of 3 months after receiving their final dose of AZD2014.
* Patient able and willing to provide informed consent with ability to understand and willingness for follow-up visits.
* Covered by a medical insurance

Exclusion Criteria:

* Patient pre-treated by a non-steroidal aromatase inhibitor
* Active uncontrolled or symptomatic central nervous system metastases or spinal cord compression
* Clinically relevant abnormal levels of potassium or sodium.
* Use of any forbidden concomitant treatment during the treatment period:

  * Any anti-cancer treatment (approved or investigational) not mentioned in the protocol
  * Chronic treatment with corticosteroids or other immunosuppressive agents. Stable low dose of corticosteroids are allowed (unless contra-indicated) provided that they were initiated before the last disease progression or were started at least 4 weeks prior to study treatment. Topical or inhaled corticosteroids are allowed.
  * Potent or moderate inhibitors or inducers of CYP3A4/5, Pgp (MDR1) and BCRP (see Appendix 5 - Restricted CYP and transporter related co-medications)
  * Sensitive or narrow therapeutic range substrates of the drug transporters OATP1B1, OATP1B3, MATE1 and MATE2K outside the wash out period and restrictions presented in Appendix 5 - Restricted CYP and transporter related co-medications)
* Patient with known hypersensitivity to anastrozole or to any of the excipients (Lactose monohydrate, Povidone, Sodium starch glycollate, Magnesium stearate, Hypromellose, Macrogol 300, Titanium dioxide)
* History of hypersensitivity to active or inactive excipients of AZD2014 or drugs with a similar chemical structure or class to AZD2014
* History of other malignancies except for basal cell or squamous cell skin cancer, in situ cervical cancer, unless they have been disease-free for at least five years
* Patient who has any severe and/or uncontrolled medical conditions such as:

  * Recent history of specific cardiovascular events, or laboratory parameters that may affect cardiac parameters including : unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to start of study drug, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease; Symptomatic congestive heart failure of New York heart Association Class III or IV
* Haemorrhagic or thrombotic stroke, including transient ischemic attack (TIA) or any other CNS bleeding.

  * Mean resting corrected QT interval (QTc), calculated using Fridericia's formula, > 470 msec obtained from 3 electrocardiograms (ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes within 12 months of the patient entering in the study
  * Abnormal cardiac function at baseline :left ventricular ejection fraction (LVEF) <50%
  * Any evidence of interstitial lung disease and uncompensated respiratory conditions.
  * Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active or chronic hepatitis (i.e. quantifiable hepatitis B virus (HBV-DNA) and/or positive HbsAg, quantifiable hepatitis C virus (HCV-RNA)),
  * Active, bleeding diathesis
  * Current refractory nausea and vomiting, chronic gastro-intestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD2014.
  * Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
  * Type 1 and uncontrolled Type 2 diabetes
  * Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with severe toxicities occurring during the first 8 weeks of follow-up assessed using National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) V4 | during the first 8 weeks of follow up
  Severe toxicities defined as
  * Any grade ≥ 4 treatment related toxicity
  * Any grade≥ 3 treatment related toxicity lasting more than 7 days
The 8-week non progression rate using RECIST v1.1 to assess tumor response to treatment | 8 weeks after start of treatment

SECONDARY OUTCOMES:
Number of patients with AE graded using CTCAE V4 | For each participant, up to 30 days after the last dose of treatment (up to 3 years)
Progression-free survival (PFS) defined as the duration of time from start of treatment to time of progression or death, whichever occurs first | up to 3 years
Overall survival (OS) defined as the duration of time from start of treatment to time of death. | 3 years
Best response rate defined as (percentage of patients with complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) according to RECIST V1.1) | Up to 3 years
Duration of objective response as per RECIST v1.1 | Up to 3 years
Area under the curve (AUC) of AZD2014 | Week 1 Day 1: pre-dose, 2h and 6-8 hours later and Week 2 Day 1: pre-dose, 2h and 6-8 hours later.
Apparent clearance of AZD2014 | Week 1 Day 1: pre-dose, 2h and 6-8 hours later and Week 2 Day 1: pre-dose, 2h and 6-8 hours later
The accumulation of the 47S precursor ribosomal ribonucleic acid (rRNA), which reflects RNA polymerase I activity analysed by fluorescence in situ hybridization (FISH) | Baseline and 8 weeks after treatment
The expression of components of rRNA methylation complex analysed by real time quantitative PCR (RTqPCR) | Baseline and 8 weeks after treatment
The levels of circulating anti-fibrillarin (anti-FBL) autoantibody on serum samples by Elisa assays | Baseline and 8 weeks after treatment
Levels of expression of fibrillarin assessed by immunohistochemistry (IHC) | Baseline and 8 weeks after treatment
Levels of expression of nucleolin assessed by IHC | Baseline and 8 weeks after treatment
Levels of expression of protein B23 assessed by IHC | Baseline and 8 weeks after treatment
Levels of expression of upstream binding factor (UBF) assessed by IHC | Baseline and 8 weeks after treatment
Levels of expression of phosphorylated UBF assessed by IHC | Baseline and 8 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Etienne HEUDEL, MD, Principal Investigator — Centre Leon Berard
Locations (12):
- France (12):
  - ICO - Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - GHM Institut Daniel Hollard, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut régional du Cancer Montpellier (ICM), Montpellier
  - Hcl - Chls, Pierre-Bénite
  - ICO - René Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Bokhman JV. Two pathogenetic types of endometrial carcinoma. Gynecol Oncol. 1983 Feb;15(1):10-7. doi: 10.1016/0090-8258(83)90111-7. PMID 6822361
- [Background] Levine DA, Hoskins WJ. Update in the management of endometrial cancer. Cancer J. 2002 May-Jun;8 Suppl 1:S31-40. PMID 12075700
- [Background] Murali R, Soslow RA, Weigelt B. Classification of endometrial carcinoma: more than two types. Lancet Oncol. 2014 Jun;15(7):e268-78. doi: 10.1016/S1470-2045(13)70591-6. PMID 24872110
- [Background] Creasman WT, Odicino F, Maisonneuve P, Quinn MA, Beller U, Benedet JL, Heintz AP, Ngan HY, Pecorelli S. Carcinoma of the corpus uteri. FIGO 26th Annual Report on the Results of Treatment in Gynecological Cancer. Int J Gynaecol Obstet. 2006 Nov;95 Suppl 1:S105-43. doi: 10.1016/S0020-7292(06)60031-3. No abstract available. PMID 17161155
- [Background] Sonoda Y. Optimal therapy and management of endometrial cancer. Expert Rev Anticancer Ther. 2003 Feb;3(1):37-47. doi: 10.1586/14737140.3.1.37. PMID 12597348
- [Background] Decruze SB, Green JA. Hormone therapy in advanced and recurrent endometrial cancer: a systematic review. Int J Gynecol Cancer. 2007 Sep-Oct;17(5):964-78. doi: 10.1111/j.1525-1438.2007.00897.x. Epub 2007 Apr 18. PMID 17442022
- [Background] Kokka F, Brockbank E, Oram D, Gallagher C, Bryant A. Hormonal therapy in advanced or recurrent endometrial cancer. Cochrane Database Syst Rev. 2010 Dec 8;2010(12):CD007926. doi: 10.1002/14651858.CD007926.pub2. PMID 21154390
- [Background] Rose PG, Brunetto VL, VanLe L, Bell J, Walker JL, Lee RB. A phase II trial of anastrozole in advanced recurrent or persistent endometrial carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2000 Aug;78(2):212-6. doi: 10.1006/gyno.2000.5865. PMID 10926805
- [Background] Diaz-Padilla I, Duran I, Clarke BA, Oza AM. Biologic rationale and clinical activity of mTOR inhibitors in gynecological cancer. Cancer Treat Rev. 2012 Oct;38(6):767-75. doi: 10.1016/j.ctrv.2012.02.001. Epub 2012 Feb 29. PMID 22381585
- [Background] Slomovitz BM, Coleman RL. The PI3K/AKT/mTOR pathway as a therapeutic target in endometrial cancer. Clin Cancer Res. 2012 Nov 1;18(21):5856-64. doi: 10.1158/1078-0432.CCR-12-0662. Epub 2012 Oct 18. PMID 23082003
- [Background] Oza AM, Elit L, Tsao MS, Kamel-Reid S, Biagi J, Provencher DM, Gotlieb WH, Hoskins PJ, Ghatage P, Tonkin KS, Mackay HJ, Mazurka J, Sederias J, Ivy P, Dancey JE, Eisenhauer EA. Phase II study of temsirolimus in women with recurrent or metastatic endometrial cancer: a trial of the NCIC Clinical Trials Group. J Clin Oncol. 2011 Aug 20;29(24):3278-85. doi: 10.1200/JCO.2010.34.1578. Epub 2011 Jul 25. PMID 21788564
- [Background] Slomovitz BM, Jiang Y, Yates MS, Soliman PT, Johnston T, Nowakowski M, Levenback C, Zhang Q, Ring K, Munsell MF, Gershenson DM, Lu KH, Coleman RL. Phase II study of everolimus and letrozole in patients with recurrent endometrial carcinoma. J Clin Oncol. 2015 Mar 10;33(8):930-6. doi: 10.1200/JCO.2014.58.3401. Epub 2015 Jan 26. PMID 25624430
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Trimble EL, Harlan LC, Clegg LX, Stevens JL. Pre-operative imaging, surgery and adjuvant therapy for women diagnosed with cancer of the corpus uteri in community practice in the United States. Gynecol Oncol. 2005 Mar;96(3):741-8. doi: 10.1016/j.ygyno.2004.11.041. PMID 15721420
- [Background] Setiawan VW, Yang HP, Pike MC, McCann SE, Yu H, Xiang YB, Wolk A, Wentzensen N, Weiss NS, Webb PM, van den Brandt PA, van de Vijver K, Thompson PJ; Australian National Endometrial Cancer Study Group; Strom BL, Spurdle AB, Soslow RA, Shu XO, Schairer C, Sacerdote C, Rohan TE, Robien K, Risch HA, Ricceri F, Rebbeck TR, Rastogi R, Prescott J, Polidoro S, Park Y, Olson SH, Moysich KB, Miller AB, McCullough ML, Matsuno RK, Magliocco AM, Lurie G, Lu L, Lissowska J, Liang X, Lacey JV Jr, Kolonel LN, Henderson BE, Hankinson SE, Hakansson N, Goodman MT, Gaudet MM, Garcia-Closas M, Friedenreich CM, Freudenheim JL, Doherty J, De Vivo I, Courneya KS, Cook LS, Chen C, Cerhan JR, Cai H, Brinton LA, Bernstein L, Anderson KE, Anton-Culver H, Schouten LJ, Horn-Ross PL. Type I and II endometrial cancers: have they different risk factors? J Clin Oncol. 2013 Jul 10;31(20):2607-18. doi: 10.1200/JCO.2012.48.2596. Epub 2013 Jun 3. PMID 23733771
- [Background] Singh M, Zaino RJ, Filiaci VJ, Leslie KK. Relationship of estrogen and progesterone receptors to clinical outcome in metastatic endometrial carcinoma: a Gynecologic Oncology Group Study. Gynecol Oncol. 2007 Aug;106(2):325-33. doi: 10.1016/j.ygyno.2007.03.042. Epub 2007 May 25. PMID 17532033
- [Background] Kauppila A. Progestin therapy of endometrial, breast and ovarian carcinoma. A review of clinical observations. Acta Obstet Gynecol Scand. 1984;63(5):441-50. doi: 10.3109/00016348409156700. PMID 6238499
- [Background] Lentz SS, Brady MF, Major FJ, Reid GC, Soper JT. High-dose megestrol acetate in advanced or recurrent endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 1996 Feb;14(2):357-61. doi: 10.1200/JCO.1996.14.2.357. PMID 8636744
- [Background] Thigpen JT, Brady MF, Alvarez RD, Adelson MD, Homesley HD, Manetta A, Soper JT, Given FT. Oral medroxyprogesterone acetate in the treatment of advanced or recurrent endometrial carcinoma: a dose-response study by the Gynecologic Oncology Group. J Clin Oncol. 1999 Jun;17(6):1736-44. doi: 10.1200/JCO.1999.17.6.1736. PMID 10561210
- [Background] Whitney CW, Brunetto VL, Zaino RJ, Lentz SS, Sorosky J, Armstrong DK, Lee RB; Gynecologic Oncology Group study. Phase II study of medroxyprogesterone acetate plus tamoxifen in advanced endometrial carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2004 Jan;92(1):4-9. doi: 10.1016/j.ygyno.2003.09.018. PMID 14751130
- [Background] Thigpen T, Brady MF, Homesley HD, Soper JT, Bell J. Tamoxifen in the treatment of advanced or recurrent endometrial carcinoma: a Gynecologic Oncology Group study. J Clin Oncol. 2001 Jan 15;19(2):364-7. doi: 10.1200/JCO.2001.19.2.364. PMID 11208827
- [Background] Ma BB, Oza A, Eisenhauer E, Stanimir G, Carey M, Chapman W, Latta E, Sidhu K, Powers J, Walsh W, Fyles A. The activity of letrozole in patients with advanced or recurrent endometrial cancer and correlation with biological markers--a study of the National Cancer Institute of Canada Clinical Trials Group. Int J Gynecol Cancer. 2004 Jul-Aug;14(4):650-8. doi: 10.1111/j.1048-891X.2004.14419.x. PMID 15304161
- [Background] Laplante M, Sabatini DM. mTOR signaling in growth control and disease. Cell. 2012 Apr 13;149(2):274-93. doi: 10.1016/j.cell.2012.03.017. PMID 22500797
- [Background] Baselga J, Campone M, Piccart M, Burris HA 3rd, Rugo HS, Sahmoud T, Noguchi S, Gnant M, Pritchard KI, Lebrun F, Beck JT, Ito Y, Yardley D, Deleu I, Perez A, Bachelot T, Vittori L, Xu Z, Mukhopadhyay P, Lebwohl D, Hortobagyi GN. Everolimus in postmenopausal hormone-receptor-positive advanced breast cancer. N Engl J Med. 2012 Feb 9;366(6):520-9. doi: 10.1056/NEJMoa1109653. Epub 2011 Dec 7. PMID 22149876
- [Background] Turina M, Christ-Crain M, Polk HC Jr. Diabetes and hyperglycemia: strict glycemic control. Crit Care Med. 2006 Sep;34(9 Suppl):S291-300. doi: 10.1097/01.CCM.0000231887.84751.04. PMID 16917434
- [Background] White DA, Camus P, Endo M, Escudier B, Calvo E, Akaza H, Uemura H, Kpamegan E, Kay A, Robson M, Ravaud A, Motzer RJ. Noninfectious pneumonitis after everolimus therapy for advanced renal cell carcinoma. Am J Respir Crit Care Med. 2010 Aug 1;182(3):396-403. doi: 10.1164/rccm.200911-1720OC. Epub 2010 Mar 1. PMID 20194812
- [Background] Albiges L, Chamming's F, Duclos B, Stern M, Motzer RJ, Ravaud A, Camus P. Incidence and management of mTOR inhibitor-associated pneumonitis in patients with metastatic renal cell carcinoma. Ann Oncol. 2012 Aug;23(8):1943-1953. doi: 10.1093/annonc/mds115. Epub 2012 Jun 11. PMID 22689175
- [Background] Ruggero D. Translational control in cancer etiology. Cold Spring Harb Perspect Biol. 2013 Feb 1;5(2):a012336. doi: 10.1101/cshperspect.a012336. PMID 22767671
- [Background] Elagoz S, Arici DS, Aker H. Relationship between FIGO grade and AgNOR, S100-positive langerhans cells in endometrial adenocarcinoma. Pathol Int. 2000 Aug;50(8):616-9. doi: 10.1046/j.1440-1827.2000.01099.x. PMID 10972859
- [Background] Trere D, Melchiorri C, Chieco P, Marabini A, Derenzini M. Interphase AgNOR quantity and DNA content in endometrial adenocarcinoma. Gynecol Oncol. 1994 May;53(2):202-7. doi: 10.1006/gyno.1994.1116. PMID 8188080
- [Background] Giuffre G, Fulcheri E, Gualco M, Fedele F, Tuccari G. Standardized AgNOR analysis as a prognostic parameter in endometrial carcinoma, endometrioid type. Anal Quant Cytol Histol. 2001 Feb;23(1):31-9. PMID 11233741
- [Background] Belin S, Beghin A, Solano-Gonzalez E, Bezin L, Brunet-Manquat S, Textoris J, Prats AC, Mertani HC, Dumontet C, Diaz JJ. Dysregulation of ribosome biogenesis and translational capacity is associated with tumor progression of human breast cancer cells. PLoS One. 2009 Sep 25;4(9):e7147. doi: 10.1371/journal.pone.0007147. PMID 19779612
- [Background] Marcel V, Ghayad SE, Belin S, Therizols G, Morel AP, Solano-Gonzalez E, Vendrell JA, Hacot S, Mertani HC, Albaret MA, Bourdon JC, Jordan L, Thompson A, Tafer Y, Cong R, Bouvet P, Saurin JC, Catez F, Prats AC, Puisieux A, Diaz JJ. p53 acts as a safeguard of translational control by regulating fibrillarin and rRNA methylation in cancer. Cancer Cell. 2013 Sep 9;24(3):318-30. doi: 10.1016/j.ccr.2013.08.013. PMID 24029231
- [Background] Choi YW, Kim YW, Bae SM, Kwak SY, Chun HJ, Tong SY, Lee HN, Shin JC, Kim KT, Kim YJ, Ahn WS. Identification of differentially expressed genes using annealing control primer-based GeneFishing in human squamous cell cervical carcinoma. Clin Oncol (R Coll Radiol). 2007 Jun;19(5):308-18. doi: 10.1016/j.clon.2007.02.010. Epub 2007 Apr 2. PMID 17399965
- [Background] Su H, Xu T, Ganapathy S, Shadfan M, Long M, Huang TH, Thompson I, Yuan ZM. Elevated snoRNA biogenesis is essential in breast cancer. Oncogene. 2014 Mar 13;33(11):1348-58. doi: 10.1038/onc.2013.89. Epub 2013 Apr 1. PMID 23542174
- [Background] Hein N, Hannan KM, George AJ, Sanij E, Hannan RD. The nucleolus: an emerging target for cancer therapy. Trends Mol Med. 2013 Nov;19(11):643-54. doi: 10.1016/j.molmed.2013.07.005. Epub 2013 Aug 15. PMID 23953479
- [Background] Burger K, Muhl B, Harasim T, Rohrmoser M, Malamoussi A, Orban M, Kellner M, Gruber-Eber A, Kremmer E, Holzel M, Eick D. Chemotherapeutic drugs inhibit ribosome biogenesis at various levels. J Biol Chem. 2010 Apr 16;285(16):12416-25. doi: 10.1074/jbc.M109.074211. Epub 2010 Feb 16. PMID 20159984
- [Background] Bywater MJ, Poortinga G, Sanij E, Hein N, Peck A, Cullinane C, Wall M, Cluse L, Drygin D, Anderes K, Huser N, Proffitt C, Bliesath J, Haddach M, Schwaebe MK, Ryckman DM, Rice WG, Schmitt C, Lowe SW, Johnstone RW, Pearson RB, McArthur GA, Hannan RD. Inhibition of RNA polymerase I as a therapeutic strategy to promote cancer-specific activation of p53. Cancer Cell. 2012 Jul 10;22(1):51-65. doi: 10.1016/j.ccr.2012.05.019. PMID 22789538
- [Background] Silvera D, Formenti SC, Schneider RJ. Translational control in cancer. Nat Rev Cancer. 2010 Apr;10(4):254-66. doi: 10.1038/nrc2824. PMID 20332778
- [Background] Hannan KM, Brandenburger Y, Jenkins A, Sharkey K, Cavanaugh A, Rothblum L, Moss T, Poortinga G, McArthur GA, Pearson RB, Hannan RD. mTOR-dependent regulation of ribosomal gene transcription requires S6K1 and is mediated by phosphorylation of the carboxy-terminal activation domain of the nucleolar transcription factor UBF. Mol Cell Biol. 2003 Dec;23(23):8862-77. doi: 10.1128/MCB.23.23.8862-8877.2003. PMID 14612424
- [Background] Iadevaia V, Liu R, Proud CG. mTORC1 signaling controls multiple steps in ribosome biogenesis. Semin Cell Dev Biol. 2014 Dec;36:113-20. doi: 10.1016/j.semcdb.2014.08.004. Epub 2014 Aug 19. PMID 25148809
- [Background] Peltonen K, Colis L, Liu H, Trivedi R, Moubarek MS, Moore HM, Bai B, Rudek MA, Bieberich CJ, Laiho M. A targeting modality for destruction of RNA polymerase I that possesses anticancer activity. Cancer Cell. 2014 Jan 13;25(1):77-90. doi: 10.1016/j.ccr.2013.12.009. PMID 24434211
- [Background] Woiwode A, Johnson SA, Zhong S, Zhang C, Roeder RG, Teichmann M, Johnson DL. PTEN represses RNA polymerase III-dependent transcription by targeting the TFIIIB complex. Mol Cell Biol. 2008 Jun;28(12):4204-14. doi: 10.1128/MCB.01912-07. Epub 2008 Apr 7. PMID 18391023
- [Background] Whittaker S, Martin M, Marais R. All roads lead to the ribosome. Cancer Cell. 2010 Jul 13;18(1):5-6. doi: 10.1016/j.ccr.2010.06.008. PMID 20609347
- [Background] Crowley E, Di Nicolantonio F, Loupakis F, Bardelli A. Liquid biopsy: monitoring cancer-genetics in the blood. Nat Rev Clin Oncol. 2013 Aug;10(8):472-84. doi: 10.1038/nrclinonc.2013.110. Epub 2013 Jul 9. PMID 23836314
- [Background] Dawson SJ, Rosenfeld N, Caldas C. Circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Jul 4;369(1):93-4. doi: 10.1056/NEJMc1306040. No abstract available. PMID 23822788
- [Background] Murtaza M, Dawson SJ, Tsui DW, Gale D, Forshew T, Piskorz AM, Parkinson C, Chin SF, Kingsbury Z, Wong AS, Marass F, Humphray S, Hadfield J, Bentley D, Chin TM, Brenton JD, Caldas C, Rosenfeld N. Non-invasive analysis of acquired resistance to cancer therapy by sequencing of plasma DNA. Nature. 2013 May 2;497(7447):108-12. doi: 10.1038/nature12065. Epub 2013 Apr 7. PMID 23563269
- [Background] Frenel JS, Carreira S, Goodall J, Roda D, Perez-Lopez R, Tunariu N, Riisnaes R, Miranda S, Figueiredo I, Nava-Rodrigues D, Smith A, Leux C, Garcia-Murillas I, Ferraldeschi R, Lorente D, Mateo J, Ong M, Yap TA, Banerji U, Gasi Tandefelt D, Turner N, Attard G, de Bono JS. Serial Next-Generation Sequencing of Circulating Cell-Free DNA Evaluating Tumor Clone Response To Molecularly Targeted Drug Administration. Clin Cancer Res. 2015 Oct 15;21(20):4586-96. doi: 10.1158/1078-0432.CCR-15-0584. Epub 2015 Jun 17. PMID 26085511
- [Derived] Heudel P, Frenel JS, Dalban C, Bazan F, Joly F, Arnaud A, Abdeddaim C, Chevalier-Place A, Augereau P, Pautier P, Chakiba C, You B, Lancry-Lecomte L, Garin G, Marcel V, Diaz JJ, Treilleux I, Perol D, Fabbro M, Ray-Coquard I. Safety and Efficacy of the mTOR Inhibitor, Vistusertib, Combined With Anastrozole in Patients With Hormone Receptor-Positive Recurrent or Metastatic Endometrial Cancer: The VICTORIA Multicenter, Open-label, Phase 1/2 Randomized Clinical Trial. JAMA Oncol. 2022 Jul 1;8(7):1001-1009. doi: 10.1001/jamaoncol.2022.1047. PMID 35551299
- See also: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTC AE) — http://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm#ctc_v40.